CLINICAL TRIAL: NCT01135875
Title: Human Glioblastoma Multiforme (GBM) Circulating Tumor Cells (CTCs) as Early, Less Invasive Markers of Progression and Response
Brief Title: Laboratory Study of Early Tumor Markers in the Peripheral Blood of Glioblastoma Multiforme Patients
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: CTC-01
Record Dates: First submitted 2010-05-24; First posted 2010-06-03 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Glioblastoma Multiforme; Healthy Volunteers
Keywords: GBM; Brain Tumor; Brain Neoplasm; Control; Normal Control; Volunteer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GBM Patients: GBM Patients with a histologically confirmed or suspected diagnosis of glioblastoma multiforme.
  Interventions: Other: GBM Patients
- Normal Controls: Normal Controls will be adult volunteers who identify themselves as not having been diagnosed with a glioblastoma multiforme.
  Interventions: Other: Normal Controls

INTERVENTIONS:
Other: GBM Patients — 2 teaspoons of blood will be collected during select clinic visits.
  Groups: GBM Patients
Other: Normal Controls — 2 teaspoons of blood will be collected once.
  Groups: Normal Controls

SUMMARY:
The purpose of this study is to determine if tumor cells can be detected in the blood of patients diagnosed with a brain tumor.

DETAILED DESCRIPTION:
Despite aggressive therapies, Glioblastoma Multiforme (GBM) is rapidly fatal. GBMs are increasingly recognized for occasionally metastasizing through the peripheral blood to distant locations. This research study involves the detection and novel characterization of human GBM (hGBM) circulating tumor cells (CTCs) within the peripheral blood of brain tumor patients by identifying their unique cell surface antigen profile, determining an optimal isolation protocol, and quantitatively and qualitatively reporting the yield and characteristics.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 89 years of age
* Weight of at least 110 pounds
* Able to provide informed consent for self

Exclusion Criteria:

* Patients with active malignant tumors other than GBM

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited during routine interactions with the investigators.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Identification of Human GBM CD Antigen Signature. | 3 Years
  Already established and stored GBM cell lines will be screened for CD antigens to confirm that a selective cell surface antigen can be identified.

SECONDARY OUTCOMES:
Identification & Isolation of Human GBM Cells in Seeded Normal Control Human Blood. | 3 Years
  Frozen and fresh human blood will be seeded with human GBM cells from established stored GBM cell lines and subjected to antibody-based cell identification and isolation procedures.
Prospective Isolation of GBM Tumor Cells in GBM Patient Blood. | 3 Years
  Circulating tumor cells will be isolated from blood drawn from GBM patients.
Prospective Evaluation of the Routine Medical History of GBM Patients. | 3 Years
  Medical records of GBM patients will be used to determine how circulating tumor cells impact outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Reynolds, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States